CLINICAL TRIAL: NCT01316835
Title: A Retrospective, Observational Study to Assess the Effectiveness of Glycemic Control of Diabetes in Real World After Sitagliptin Usage
Brief Title: Effectiveness of Sitagliptin in Glycemic Control in Real World
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Ching-Jung Hsieh/ Head of department, Chang Gung Memorial Hospital
Other Study IDs: 99-2717B
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: retrospective,sitagliptin, glycemia control,real world
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus, No treatment

SUMMARY:
This study will evaluate whether the addition of sitagliptin treatment provides additional decrease in HbA1C levels and increase in goal attainment in patients with inadequate glycemic control on their current oral anti-glycemic therapy in real world practice.

DETAILED DESCRIPTION:
To explore the change of glycemic control (HbA1c or FPG) before and after 24 weeks of Sitagliptin treatment in Type 2 Diabetic patients who have started Sitagliptin as add on therapy during the index period and received Sitagliptin continuously* for at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects diagnosed of type 2 diabetes (ICD-9 code= 250.0; 250.1; 250.2; 250.3; 250.4; 250.5; 250.6) and have been followed up regularly in the study center who have started to receive Sitagliptin as an add-on treatment to their prior regimen during the index period
2. Subjects must be on a stable dose of all antidiabetic regimens, with stable dose defined as "at least 3 months with no therapy/dose change" prior to adding sitagliptin
3. Subjects in whose medical records a minimum core data set can be found.
4. Outpatient

Exclusion Criteria:

1. Subjects with type 1 DM
2. Subjects have been treated with insulin regularly
3. Subject with DM which results from other general diseases, e.g. surgery, pharmaceutical products, malnutrition, infections and other conditions
4. Subjects who participated in a clinical trial or other clinical study during the index period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with ICD-9 diagnostic codes of T2DM plus any prescription record of the anti-glycemic drugs included in the hospital formulary during the study period will be extracted from the hospital outpatient electronic database. Sitagliptin users who stayed with Sitagliptin for at least 24 weeks will then further identified from this diabetes cohort for efficacy analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Jung Hsieh, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospita, Kaohsiung City, Taiwan